CLINICAL TRIAL: NCT06703073
Title: Phase 2 Clinical Platform Trial Investigating Multiple Therapeutic Options for the Treatment of Hospitalized Patients With Acute Respiratory Distress Syndrome (ARDS)
Brief Title: JUST BREATHE, Breathing Life Into Innovative Therapies for ARDS (Master Record)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PPD Development, LP (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); InflaRx GmbH (Industry); Edesa Biotech Inc. (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BP-ARDS-P2-001 (Master Record); 75A50124C00001 (Other Grant/Funding Number: Biomedical Advanced Research and Development Authority (BARDA))
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); ARDS; ARDS (Acute Respiratory Distress Syndrome); Acute Respiratory Distress Syndrome
Keywords: BARDA; JUST BREATHE; ARDS; Acute Respiratory Distress Syndrome; Acute Respiratory Failure
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The overall 2-step randomization scheme will be implemented.
  * Randomization Level 1 will be open-label, assigning an eligible patient to one of the available treatment cohorts.
  * Randomization Level 2 will be double-blinded and will randomize participants at a 1:1 ratio to receive either IP or placebo within a specific cohort. Thus, the PPD blinded team, site blinded staff members, and participants/legal authorized representative will be considered blinded to study treatment assignment (either IP or placebo) throughout the course of the study.
  To preserve the integrity of the study blind, an unblinded pharmacist at each site will be responsible for the reconstitution and dispensation of all study drugs and placebos and will endeavor to ensure that there are no observable differences between the treatment groups (IP or placebo) when dispensing the study materials.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort A: vilobelimab (Experimental)
  Interventions: Drug: Cohort A: vilobelimab
- Cohort A: placebo (Placebo Comparator)
  Interventions: Drug: Cohort A: placebo
- Cohort B: paridiprubart (Experimental)
  Interventions: Drug: Cohort B: paridiprubart
- Cohort B: placebo (Placebo Comparator)
  Interventions: Drug: Cohort B: placebo
- Cohort C: bevacizumab (Experimental)
  Interventions: Drug: Cohort C: bevacizumab
- Cohort C: placebo (Placebo Comparator)
  Interventions: Drug: Cohort C: placebo

INTERVENTIONS:
Drug: Cohort A: vilobelimab — Administered as an IV formulation of 800 mg per dose and up to 6 doses (planned for Days 1, 2, 4, 8, 15, and 22, if participant is in hospital setting and deemed appropriate by the investigator)
  Arms: Cohort A: vilobelimab
Drug: Cohort A: placebo — Administered as an IV formulation of placebo of up to 6 doses (planned for Days 1, 2, 4, 8, 15, and 22, if participant is in hospital setting and deemed appropriate by the investigator)
  Arms: Cohort A: placebo
Drug: Cohort B: paridiprubart — Administered as a single IV dose of 15 mg/kg up to maximum of 1440 mg on Day 1
  Arms: Cohort B: paridiprubart
Drug: Cohort B: placebo — Administered as a single IV dose of placebo on Day 1
  Arms: Cohort B: placebo
Drug: Cohort C: bevacizumab — Administered as a single IV dose of 500 mg on Day 1
  Arms: Cohort C: bevacizumab
Drug: Cohort C: placebo — Administered as a single IV dose of placebo on Day 1
  Arms: Cohort C: placebo

SUMMARY:
This is a Phase 2 multicenter, randomized, double-blinded, placebo-controlled study that will evaluate the safety and efficacy of host-directed therapeutics in hospitalized adults diagnosed with Acute Respiratory Distress Syndrome (ARDS) utilizing a platform trial design. Participants will be randomized to receive either a placebo or one of the active treatments.

This record describes the default procedures and analyses for all cohorts. Each specific cohort may have additional eligibility requirements, safety and efficacy procedures, or endpoints, which will be described in the corresponding intervention-specific records on clinicaltrials.gov listed below in the detailed description.

DETAILED DESCRIPTION:
This is a master protocol for a Phase 2 platform clinical trial to evaluate host-directed therapeutic candidates (i.e., investigational product, IP) for the treatment of hospitalized participants diagnosed with ARDS. The safety and efficacy of each IP will be studied within its own cohort (IP versus Placebo). All patients will continue to receive standard treatments for ARDS as per the investigator. An individual participant will complete the study in approximately 90 days. The study will include a screening period (<24 hours from providing informed consent to treatment), in-hospital treatment period with IP/placebo starting on Day 1 through discharge from the hospital, and a follow-up period after discharge from the hospital through the end of study (Day 90 + 2 weeks).

Outcome data will be assembled for each patient over time (such as ventilatory status, oxygenation, and survival). Functional status using the WHO Ordinal scale and Karnofsky scale will be collected. Resource utilization will be calculated (length of stay in a critical care setting, days intubated, and survival).

All participants will undergo a series of physical exams, laboratory assessments/biomarker collections, ECG, Chest X-ray or CT scan, and questionnaires through Day 90. Exploratory biomarkers will be evaluated over time to facilitate clinical learning.

For information specific to each intervention included in this platform trial, please refer to the below corresponding, separate, clinicaltrials.gov records:

Vilobelimab NCT06701682 ; Paridiprubart NCT06701669 ; Bevacizumab NCT06701656

ELIGIBILITY:
Inclusion Criteria:

* Participant (or their Legally Authorized Representative (LAR)) provides informed consent and agrees to comply with protocol requirements
* Participant is at least 18 years of age or older at the time of consent.
* Participant with signs and symptoms of ARDS according to the Berlin definition of ARDS.

Note that participants on noninvasive ventilation may be screened.

* Participant of childbearing potential must agree to either abstinence or use at least one primary form of contraception, not including hormonal contraception, from the time of screening through Day 28. Additional cohort-specific requirements may apply
* Participant agrees to not participate in another investigational interventional study while participating in this study (i.e., through Day 90).

Exclusion Criteria:

* Participant with ARDS or at risk of developing ARDS due to the following reasons: trauma, large volume aspiration, or transfusion.
* Participant with pulmonary edema due to cardiogenic pulmonary edema/fluid overload or hypoxemia primarily attributable atelectasis, in the absence of a predisposing risk factor for ARDS.
* Participant who demonstrates an improvement in oxygenation and ventilatory support 24 hours prior to or during screening up to randomization, such that per investigator clinical judgement, the participant is expected to have significant improvement in lung function over subsequent 24 hours regardless of additional interventions.
* Participant is known to be pregnant, nursing, or with a positive (urine and/or serum test) pregnancy test.
* Participant is anticipated to be transferred to another hospital which is not a study site within 72 hours.
* Participant is not expected to survive for 72 hours.
* Participant has been on invasive mechanical ventilation or ECMO for more than 48 hours for ARDS at the time of consent.
* Participant has an underlying clinical condition where, in the opinion of the Investigator and based on their clinical judgement, it would be extremely unlikely that the participant would come off ventilation
* Participant has severe COPD requiring continuous long-term home oxygen therapy or mechanical ventilation (noninvasive ventilation or via tracheotomy) except for CPAP or bi-level positive airway pressure used solely for sleep-disordered breathing.
* Participant has interstitial lung disease or idiopathic pulmonary fibrosis requiring continuous chronic home oxygen therapy.
* Participant has NY Heart Association Class IV congestive heart failure.
* Participant has a known allergy to any study medication or any of its excipients.
* Participant is receiving systemic immunosuppressive therapy for solid organ or hematopoietic cancer or transplant anti-rejection medication.

NOTE: Patients on chronic low dose immunosuppressive therapy may be enrolled at the discretion of the investigator in consultation with the medical monitor.

* Participant is undergoing active cancer systemic chemotherapy.
* Participant received treatment with an investigational immunomodulator or immunosuppressant drugs within 5 half-lives or 30 days (whichever is longer) before randomization.
* Participant with concurrent infections or history of the following:

  1. Known active tuberculosis,
  2. Known active Hepatitis B, or
  3. HIV and a CD4 count less than 50 or a detectable viral load of >200 copies/mL HIV RNA.
* Participant received treatment with any other investigational drugs within 30 days prior to consent.
* Participant had a history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess within 28 days of screening or inadequate wound healing secondary to major thoracoabdominal surgery at the time of screening.
* Participant is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Participant may have additional cohort-specific requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality (ACM) rate at Day 28 | Day 28

SECONDARY OUTCOMES:
ACM at Day 60 and Day 90 | Day 60 and Day 90
ACM+ at Day 28, Day 60, and Day 90 | Day 28, Day 60, and Day 90
  Note: ACM+ composite score will be constructed by combining ACM and participant-relevant, infection-related Adverse Events (AE) from the MedDRA toxic/septic shock standardized MedDRA queries.
Improvements in oxygenation measured as change from baseline in PaO2/FiO2 ratio up to and including Day 28 (or discharge, whichever is earlier) | Up to and including Day 28 or until Discharge (whichever is earlier)
Incidence of new invasive mechanical ventilation use during the study up to and including Day 28 | Up to and including Day 28
Ventilator-free days up to and including Day 28 | Up to and including Day 28
Proportion of participants alive and free of mechanical ventilation at Days 28, 60, and 90 | Days 28, 60, and 90
Time to recover gas exchange to a PaO2/FiO2 ≥ 300 measured on 2 consecutive days during the first 28 days after informed consent | Up to and including Day 28
Extracorporeal Membrane Oxygenation (ECMO) free days up to and including Day 28 | up to and including Day 28
Incidence of participants with new ECMO use during the study up to and including Day 28. | up to and including Day 28
Proportion of participants alive and free of ECMO at Days 28, 60, and 90 | Days 28, 60, and 90.
Proportion of participants achieving a ≥2-point improvement from baseline in the World Health Organization (WHO) 8-levels ordinal scale (from 0-8) | While Hospitalized (up to 90 days)
Time to an improvement of one category and two categories from baseline using the WHO 8-levels ordinal scale (from 0-8) at Days 28, 60, and 90 (while hospitalized) | While Hospitalized (up to 90 days)
Mean change in the WHO 8-levels ordinal scale from baseline through Day 90 (while hospitalized) | While Hospitalized (up to 90 days)
Proportion of participants who improve clinical status as measured by the Karnofsky scale | Post hospitalization through Day 90
  The Karnofsky scale is used to assess the general condition of the patient. Scores range from 0 to 100 with higher scores indicating better functional ability.
Days of hospitalization up to and including Day 28 | up to and including Day 28
Days of ICU stay up to and including Day 28 | up to and including Day 28
Change in Short Form Health Survey (SF-12) from hospital discharge to Day 60 and to Day 90 | From hospital discharge to Day 60 and to Day 90
  The SF-12 is a self-reported outcome measure composed by 12 items which examine eight dimensions of physical and mental health. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Change in St. George's Respiratory Questionnaire (SGRQ) from hospital discharge to Day 60 and to Day 90 | From hospital discharge to Day 60 and to Day 90
  The SGRQ comprises of 50 items and consists of two parts. The first part pertains to symptoms and the second pertains to functional status as well as social and psychological impact of disease. Overall scores range between 0 and 100 with higher scores indicating more limitations.
Incidence and severity of adverse events (AEs) /adverse event of special interest (AESI) / serious adverse event (SAEs) | Through Day 90

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Community Regional Medical Center, Fresno, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - University of California Irvine Medical Center, Orange, California
  - University of California Davis Medical Center - Pulmonary Medicine, Sacramento, California
  - Denver Health Hospital and Authority, Denver, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Nova Clinical Research, Bradenton, Florida
  - North Florida / South Georgia Veterans Health System, Gainesville, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - St. Luke's Boise Medical Center, Boise, Idaho
  - OSF Saint Francis Medical Center-, Peoria, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Henry Ford Health Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Renown Institute for Heart & Vascular Health, Reno, Nevada
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Montefiore Hospital - Moses Campus, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Mercy Health - St. Vincent Medical Center, Toledo, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Truwit JD, Fleming K, Nanchal RS. Empowering Respiratory Therapists to Restrict Nebulized 3% Saline and N-Acetylcysteine During Mechanical Ventilation. Respir Care. 2025 Aug;70(8):937-945. doi: 10.1089/respcare.12586. Epub 2025 Feb 24. PMID 40028879